CLINICAL TRIAL: NCT07096245
Title: Conectados: Social Networks and Social Media for Vaccine Uptake
Acronym: Conectados
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-38709
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Vaccination
Keywords: vaccination; social media; intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social media (Active Comparator): Participants in this arm will view a short (2-3 minute) educational video about flu and COVID-19 vaccines through paid advertisements on Facebook and Instagram. After viewing the video, they will be asked to respond to a single poll question: "How much do you trust this video?" Participants will then be invited to complete an optional, anonymous online survey assessing vaccine confidence, trust in the information source, and willingness to share the video. All procedures are self-directed and occur online.
  Interventions: Behavioral: Vaccine Information Video Dissemination
- Participant seed (Experimental): Participants in this arm are individuals who previously completed a related survey and consented to be recontacted. These "seed" participants receive a personalized video link and instructions to share it with at least 10 people in their personal networks. They will first watch the same 2-3 minute vaccine education video, answer a 1-question poll ("How much do you trust this video?"), and complete an anonymous online survey assessing vaccine attitudes, trust in the message and source, and willingness to share. Recipients of their shared video link may also complete the poll and survey. Sharing patterns are tracked via unique link analytics.
  Interventions: Behavioral: Vaccine Information Video Dissemination
- Community based organizations (Experimental): Participants in this arm will view a short educational video about flu and COVID-19 vaccines distributed by trusted community-based organizations (CBOs) using their usual communication methods, such as WhatsApp, email, newsletters, or social media. After watching the video, participants will be asked to answer a 1-question poll ("How much do you trust this video?") and will be invited to complete an optional, anonymous online survey assessing vaccine attitudes, trust in the source of the information, and willingness to share the video. CBOs will use unique tracking links to monitor video engagement.
  Interventions: Behavioral: Vaccine Information Video Dissemination

INTERVENTIONS:
Behavioral: Vaccine Information Video Dissemination — The intervention is a brief, community-informed educational video (2-3 minutes) focused on seasonal flu and COVID-19 vaccination. The video was developed using human-centered design and community-based participatory methods with Indigenous community members in California. It aims to promote trust in vaccines by presenting clear, culturally relevant health information.
  The video is disseminated using three behavioral delivery strategies: (1) paid advertisements on Facebook and Instagram targeting adults in California, (2) peer-to-peer sharing by participants who previously enrolled in the study and are invited to serve as "seeds" who share the video with their personal contacts, and (3) distribution by trusted community-based organizations (CBOs) using their existing communication networks, including WhatsApp, social media, email, and newsletters. All viewers are prompted to complete a one-question trust poll and invited to participate in an optional anonymous survey on vaccine attitud

SUMMARY:
This study is testing different ways of sharing a short, community-informed video about flu and COVID-19 vaccines to see how people respond to it. The video was created with input from Indigenous community members in California and provides information to support vaccine decision-making. Participants may see the video in one of three ways: through a paid advertisement on social media, from a trusted community organization, or from someone they know personally. After watching the video, viewers will be asked to answer one question about how much they trust it, and they may choose to complete a short survey about their vaccine views and how they received the video. The goal is to understand how trust in vaccine information changes depending on who shares it, and to improve the way health messages are delivered to Indigenous and other underserved communities.

DETAILED DESCRIPTION:
This is a randomized dissemination trial evaluating the impact of different message delivery strategies on trust, attitudes, and behavioral intentions related to flu and COVID-19 vaccination. The intervention consists of a short (approximately 2-minute) culturally tailored video, developed using human-centered design and community-based participatory approaches with Indigenous communities in California.

Participants are exposed to the video through one of three dissemination arms: (1) paid advertisements on Facebook and Instagram targeting adults 65 and older in California; (2) peer-to-peer sharing by "seed" participants recruited from a prior phase of the study; and (3) community-based organization (CBO) outreach using established communication channels. All participants view the same video.

After viewing the video, participants are asked to respond to a single poll item ("How much do you trust this video?") and are invited to complete an optional, anonymous online survey assessing vaccine confidence, trust in the information source, and willingness to share the video. Survey responses are linked to the dissemination arm for comparative analysis.

Seed participants receive personalized, trackable video links and instructions to share them with at least 10 contacts in their network. Click-level analytics (e.g., timestamp, referral source, general location) are collected through Bitly or Rebrandly links. YouTube analytics will also be used to evaluate video engagement (e.g., views, retention, traffic source). No identifiable health information is collected unless participants voluntarily provide contact information to complete the survey by phone.

The primary outcome is the level of trust in the video across dissemination arms. Secondary outcomes include survey completion rate, willingness to share the video, and changes in vaccine-related attitudes. Data will be stratified by dissemination method and, for seed participants, linked to prior social network data collected in Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Currently resides in California
* Able to access and view an online video
* Able to complete an online survey in English or Spanish For Arm 2 only (Participant Seed Arm): must have participated in the prior Aim 1 survey and consented to recontact

Exclusion Criteria:

* Under 18 years of age
* Does not reside in California
* Unable to access the internet to view the intervention video or complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Trust in vaccine video message by dissemination arm | immediately after exposure
  Participants will be asked to answer a single poll question after viewing a 2-3 minute vaccine education video: "How much do you trust this video?" Responses will be collected on a 4-point Likert scale (Not at all, A little, Mostly, Completely). The primary outcome is the level of trust reported, compared across dissemination arms (paid social media ads, peer-to-peer sharing, and community-based organization distribution). Analysis will assess differences in trust levels based on who shared the video.
Intention | Immediately after video exposure
  Assesses participants' reported likelihood of getting a seasonal flu or COVID-19 vaccine after viewing the intervention video. Measured on a 6-point scale from "Very unlikely" to "Very likely," including an option for participants who have already received the vaccine. Analysis will examine variation by dissemination arm and correlation with trust in the video.

SECONDARY OUTCOMES:
Self-reported exposure to new information | Immediately after video exposure
  Participants are asked whether the video provided them with new information related to flu or COVID-19 vaccines. This binary outcome (Yes/No/Not sure) helps assess the video's educational value.
Trust in message source | Immediately after video exposure
  Assesses how much participants trust the person or group from whom they received the video. Measured on a 4-point scale (Not at all, A little, Mostly, Completely).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual-level survey data collected through the optional online Qualtrics survey, including participants' self-reported trust in the video, vaccine attitudes, exposure history, sharing behavior, and demographics (e.g., age group, gender, Indigenous identification). No names, contact information, or IP addresses will be shared. Data will be available to qualified researchers upon reasonable request and subject to data use agreements that protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF